CLINICAL TRIAL: NCT06135064
Title: Deep Brain Therapy With Low-intensity Ultrasound for Treatment of Post-traumatic Stress Disorder
Brief Title: Ultrasonic Neuromodulation for Treatment of PTSD
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: IRB administrative closure
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Jan Kubanek, Assistant Professor, University of Utah
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB_00173062
Record Dates: First submitted 2023-11-08; First posted 2023-11-18 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-04

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active stimulation (Experimental): Low-intensity transcranial focused ultrasound stimulation of deep brain targets affected by PTSD.
  Interventions: Device: Diadem
- Sham stimulation (Sham Comparator): Sham stimulation that applies the device in the same way as verum but only delivers auditory sounds correspoding to the ultrasonic pulses.
  Interventions: Device: Diadem

INTERVENTIONS:
Device: Diadem — The device delivers low-intensity ultrasonic waves into specified brain targets.

SUMMARY:
This study will evaluate a new form of non-invasive deep brain therapy for individuals with post-traumatic stress disorder (PTSD). Low-intensity transcranial focused ultrasound stimulation will first be delivered using a range of stimulation parameters during psychophysical and physiological monitoring. A well-tolerated stimulation protocol will be selected for subsequent testing in a blinded randomized sham-controlled cross-over trial. The trial will evaluate brain target engagement using magnetic resonance imaging and numerical scales of PTSD, cognitive performance, and mood.

ELIGIBILITY:
Inclusion Criteria:

* Positive PTSD diagnosis; PCL-5 > 20

Exclusion Criteria:

* Inability to complete MRI
* Suicidal ideation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-04-05 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | Up to 3 months following study initiation
  20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. The total severity scores range from 0 to 80.

SECONDARY OUTCOMES:
National Institutes of Health Toolbox Cognitive Battery (NIHTB-CB) | Up to 3 months following study initiation
  The NIHTB-CB provides the following summary scores: Total Cognition Composite, Fluid Composite (includes Dimensional Change Card Sort, Flanker Inhibitory Control and Attention, Picture Sequence Memory (Form A), List Sorting Working Memory, and Pattern Comparison tests), and Crystallized Composite (includes Picture Vocabulary and Oral Reading Recognition tests). The scores are normalized to have a mean score of 10 and standard deviation of 3.
California Verbal Learning Test, 3rd Edition (CVLT3) | Up to 3 months following study initiation
  A verbal learning and memory test designed to test immediate recall, short delay recall, long delay recall, and recognition memory, as well as the memory strategies being used by the participant. The Brief Form of the CVLT 3 consists of nine words, administered repeatedly over 4 immediate recall trials. The scoring software provides normative data.
PROMIS scale of Pain Intensity | Up to 3 months following study initiation
  The score assess the worst, average, and current levels of pain on a scale from 1 (no pain) to 5 (very severe)
Hamilton Depression Rating Scale (HDRS-17) | Up to 3 months following study initiation
  This 17-item questionnaire rates the severity of depression by probing mood, feelings of guilt, suicide ideation, insomnia, agitation or retardation, anxiety, weight loss, and somatic symptoms. The scores range from 0 (no symptoms) to 52 (worst possible).
Pittsburgh Sleep Quality Index (PSQI) | Up to 3 months following study initiation
  Test consisting of 7 components summed to yield a global PSQI score, ranging from of 0 (good sleep) to 21 (poor sleep).

CONTACTS AND LOCATIONS:
Overall Officials: Jan Kubanek, PhD, Principal Investigator — University of Utah; Elisabeth Wilde, PhD, Study Chair — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No